CLINICAL TRIAL: NCT04144244
Title: Comparison of the Effect of Microfluid Sperm Sorting Chip and Density Gradient Methods on Pregnancy Success in Intrauterine Insemination Cycles ; a Randomised Controlled Study
Brief Title: Comparison of the Effect of Microchip and Density Gradient Methods in Intrauterine Insemination Cycles
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Microchip IUI study
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Infertility Unexplained; Infertility, Male
Keywords: microfluid chip; gradient-density; intrauterine insemination
MeSH Terms: conditions — Infertility, Male | interventions — Centrifugation, Density Gradient

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MicroFluidic Sperm Sorting Chips (Experimental): Sperm Sorting microfluidic chips will be used when preparing sperm of male partner and IUI will be made with separated sperm
  Interventions: Other: MicroFluidic Sperm Sorting Chips
- gradient-density centrifugation (Active Comparator): gradient-density centrifugation technique will be used when preparing sperm of male partner and IUI will be made with separated sperm
  Interventions: Other: Gradient-Density Centrifugation

INTERVENTIONS:
Other: MicroFluidic Sperm Sorting Chips — sperm selection of IUI treatment
  Arms: MicroFluidic Sperm Sorting Chips
Other: Gradient-Density Centrifugation — sperm selection of IUI treatment
  Arms: gradient-density centrifugation

SUMMARY:
Microfluidic chips are one of the methods of sperm separation to eliminate DNA fragmentation in sperm. It is thought that the separation of sperm by centrifugation in the classical gradient density (Percoll) method used in sperm separation in IVF and IUI cycles leads to the increase of reactive oxygen radicals in sperm and this leads to sperm DNA fragmentation. Studies comparing Percoll and microfluidic chip method in terms of sperm, embryo quality and pregnancy rates are limited. In this context, it is aimed to investigate the effect of Percoll or Microfluidic Chip Technology on the quality of sperms and embryos obtained with these sperms and their pregnancy rates prospectively.

DETAILED DESCRIPTION:
The increase in infertility rate due to environmental and physiological conditions leads to an increase in the use of assisted reproductive techniques. Isolation of living and morphologically normal live sperm is an integrated procedure in commonly used IVF / ICSI(intracytoplasmic sperm injection) / IUI(intrauterine insemination) procedures. Although current IUI procedures result in a successful pregnancy of around 10-15%, the process can be greatly compromised if the selected sperm is abnormal. Microfluidic chips are one of the recommended sperm separation methods to eliminate DNA fragmentation in sperm. It is thought that the separation of the sperm by centrifugation in the classical gradient density (Percoll) method which is used in the separation of sperm in the IUI cycles, causes the increase of reactive oxygen radicals in sperm and this leads to sperm DNA fragmentation. Studies comparing Percoll and microfluidic chip method in terms of sperm, embryo quality and pregnancy rates are limited. In this context, it is aimed to investigate the effect of Percoll or Microfluidic Chip Technology on the quality of sperms and embryos obtained with these sperms and their pregnancy rates prospectively.

ELIGIBILITY:
Inclusion Criteria:

* Apply to the infertility clinic due to unexplained infertility and mild male factor (total motile sperm count >5 million)
* Volunteer

Exclusion Criteria:

* Inadequate follicle development with medication
* Embryo does not have the appropriate quality for transfer
* Tubal pathology
* Total motile sperm count < 5 million
* Refuse to participate in research

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 176 (Estimated)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-05-15 (Estimated); Study Completion 2020-07-15 (Estimated)

PRIMARY OUTCOMES:
Compare microfluid chip and density-gradient methods in terms of IUI success | average of 6 months
  measure the clinical pregnancy rate by using serum beta-HCG (human chorionic gonadotropin) level
Compare microfluid chip and density-gradient methods in terms of embryo quality | average of 6 months
  Embryo morphology will be assessed on day 3 using the standard criteria of the number of blastomeres and extent of fragmentation and blastomere asymmetry. Top quality embryos on day 3 will be designated as embryos with 7-8 cells, ≤10% fragmentation, and symmetric blastomeres. Using these criteria, the rate of top quality embryos will be analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem University, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Gode F, Bodur T, Gunturkun F, Gurbuz AS, Tamer B, Pala I, Isik AZ. Comparison of microfluid sperm sorting chip and density gradient methods for use in intrauterine insemination cycles. Fertil Steril. 2019 Nov;112(5):842-848.e1. doi: 10.1016/j.fertnstert.2019.06.037. Epub 2019 Sep 19. PMID 31543253
- [Background] Yetkinel S, Kilicdag EB, Aytac PC, Haydardedeoglu B, Simsek E, Cok T. Effects of the microfluidic chip technique in sperm selection for intracytoplasmic sperm injection for unexplained infertility: a prospective, randomized controlled trial. J Assist Reprod Genet. 2019 Mar;36(3):403-409. doi: 10.1007/s10815-018-1375-2. Epub 2018 Dec 12. PMID 30542782